CLINICAL TRIAL: NCT03278431
Title: Different Drug Combinations Against Hookworm Infection in School-aged Children in the Lao People's Democratic Republic, a Single Blind, Randomised Controlled Trial
Brief Title: Triple Combinations Against Hookworm Infections in Lao
Acronym: Tricombi
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Swiss Tropical & Public Health Institute (Other)
Responsible Party: Principal Investigator, Jennifer Keiser, Prof, Swiss Tropical & Public Health Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TRICOMBI01032017
Record Dates: First submitted 2017-09-06; First posted 2017-09-11 (Actual); Last update posted 2018-05-08 (Actual); Status verified 2018-05

CONDITIONS: Hookworm Infection
MeSH Terms: conditions — Hookworm Infections | interventions — Albendazole; Pyrantel Pamoate; oxantel pamoate; Mebendazole

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Albendazole triple combi (Active Comparator): Albendazole (400 mg) + pyrantel pamoate (20 mg/kg) + oxantel pamoate (20 mg/kg)
  Interventions: Drug: Albendazole; Drug: Pyrantel Pamoate; Drug: Oxantel Pamoate
- Pyrantel pamoate double combi (Experimental): Pyrantel pamoate (20 mg/kg) + oxantel pamoate (20 mg/kg)
  Interventions: Drug: Pyrantel Pamoate; Drug: Oxantel Pamoate
- Albendazole double combi (Experimental): Albendazole (400 mg) + oxantel pamoate (20 mg/kg)
  Interventions: Drug: Albendazole; Drug: Oxantel Pamoate
- Mebendazole triple combi (Experimental): Mebendazole (500mg) + pyrantel pamoate (20 mg/kg) + oxantel pamoate (20 mg/kg)
  Interventions: Drug: Pyrantel Pamoate; Drug: Oxantel Pamoate; Drug: Mebendazole

INTERVENTIONS:
Drug: Albendazole — Albendazole (400 mg) from Janssen, donated by the World Health Organization
  Arms: Albendazole double combi; Albendazole triple combi
Drug: Pyrantel Pamoate — Pyrantel pamoate (20 mg/kg), will be purchased by the World Health Organization
  Arms: Albendazole triple combi; Mebendazole triple combi; Pyrantel pamoate double combi
Drug: Oxantel Pamoate — Oxantel pamoate (20mg/kg) will be produced by the University of Basel
Drug: Mebendazole — Mebendazole (500 mg) from GlaxoSmithKline, donated by the World Health Organization
  Arms: Mebendazole triple combi

SUMMARY:
More than one billion people are infected with soil-transmitted helminths (STH, A. lumbricoides, hookworm or Trichuris trichiura). Preventive chemotherapy - i.e. annual or biannual treatment of at-risk populations with albendazole or mebendazole is the current strategy against STH. However, the efficacy of both drugs is only moderate against hookworm and low against T. trichiura. For increasing the efficacy and to avoid drug resistance, new drugs or the combination of different drugs is the way forward.

In this randomised controlled trial, we assess the efficacy (based on cure rates) of different drug combinations in school-aged children in Lao. 420 hookworm positive children will be treated: 140 with albendazole-oxantel pamoate, 140 with albendazole-pyrantel pamoate-oxantel pamoate treatment arms, 70 with pyrantel pamoate-oxantel pamoate and 70 with mebendazole-pyrantel pamoate-oxantel pamoate. Two stool samples will be collected at baseline and follow-up (14-21 days after treatment) and analysed with Kato-Katz.

DETAILED DESCRIPTION:
More than one billion people are infected with A. lumbricoides, hookworm or Trichuris trichiura, the so-called soil-transmitted helminths (STH). Preventive chemotherapy - i.e. annual or biannual treatment of at-risk populations, is the current strategy against STH advocated by the World Health Organization. However, the currently used drugs albendazole and mebendazole have only moderate efficacy against hookworm and low against T. trichiura. The main challenge is their temporal decrease in efficacy, which might be associated with drug resistance, as it was shown in veterinary medicine. For increasing the efficacy and to avoid drug resistance, new drugs or the combination of different drugs is the way forward.

The primary objective of this study is to assess the efficacy (based on cure rates [CR]) of the three combinations, i.e. albendazole-oxantel pamoate, pyrantel pamoate-oxantel pamoate and albendazole-pyrantel pamoate-oxantel pamoate in school-aged children infected with hookworms in Laos. Secondary objectives include; i) a proof of concept, investigating the difference between the two triple combinations albendazole-pyrantel pamoate-oxantel pamoate versus mebendazole-pyrantel pamoate-oxantel pamoate (based on CRs), ii) egg reduction rates (ERR) against hookworm and ERRs/CRs against A. lumbricoides and T. trichiura and iii) tolerability of the 4 combinations.

Two stool samples will be collected from school-aged children (age 6-15) at baseline. 420 hookworm positive children will be treated: 140 with albendazole-oxantel pamoate, 140 with albendazole-pyrantel pamoate-oxantel pamoate, 70 with pyrantel pamoate-oxantel pamoate and 70 with mebendazole-pyrantel pamoate-oxantel pamoate treatment arms The medical history of the participating children will be assessed with a standardized questionnaire, in addition to a clinical examination carried out by the study physician on the treatment day. Children will be interviewed before treatment for clinical symptoms and 3 and 24 hours after treatment about the occurrence of adverse events. The efficacy of the treatment will be determined 14-21 days post-treatment by collecting another two stool samples. All stool samples will be examined with duplicated Kato-Katz thick smears.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent signed by parents and/or legal representative; and a verbal assent (children <12 years) or signed assent (children ≥12 years), according to Lao regulations.
* Able and willing to be examined by a study physician at the beginning of the study.
* Able and willing to provide two stool samples at the beginning (baseline) and two to three weeks after treatment (follow-up).
* Positive for hookworm eggs in the stool.
* Absence of major systemic illnesses, e.g. diabetes, severe anemia as assessed by a medical doctor, upon initial clinical assessment.
* No known or reported history of chronical illness as cancer, diabetes, chronic heart, liver or renal disease.
* No recent anthelminthic treatment (within past 4 weeks).
* No known allergy to study medications (e.g. albendazole, mebendazole, pyrantel pamoate, oxantel pamoate).
* Negative pregnancy test (girls ≥12 years)

Exclusion Criteria:

* No written informed consent by parents and/or legal representative and no verbal assent (children <12 years) or signed assent (children ≥12 years).
* Presence of major systemic illnesses, e.g. diabetes, severe anemia as assessed by a medical doctor, upon initial clinical assessment.
* History of acute or severe chronic disease.
* Recent use of anthelminthic drug (within past 4 weeks).
* Attending other clinical trials during the study.
* Negative diagnostic result for hookworm eggs in the stool.
* Positive pregnancy test (girls ≥12 years)

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 420 (Actual)
Dates: Start 2017-09-27 (Actual); Primary Completion 2017-11-17 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
Cure rates of three drug combinations | 14-21 days after treatment
  to comparatively assess the efficacy (based on cure rates, CR) i) albendazole-oxantel pamoate, ii) pyrantel pamoate-oxantel pamoate, iii) albendazole-pyrantel pamoate-oxantel pamoate in school-aged children infected with hookworms.

SECONDARY OUTCOMES:
Cure rates against hookworm of the two triple combinations | 14-21 days after treatment
  To assess the CRs against hookworm of albendazole-pyrantel pamoate-oxantel pamoate versus mebendazole-pyrantel pamoate-oxantel pamoate (proof of concept)
Egg reduction rates (ERR) against hookworm and ERRs/CRs against A. lumbricoides and T. trichiura | 14-21 days after treatment
  Assessing the egg reduction rates (ERR) against hookworm and ERRs and cure rates (CR) against A. lumbricoides and T. trichiura
Incidence of adverse events 3 and 24 hours after treatment | 3 and 24 hours after treatment
  Participants will be interviewed using a standardized questionnaire, before treatment for clinical symptoms and 3 and 24 hours after treatment about the occurrence of adverse events.

CONTACTS AND LOCATIONS:
Locations (1):
- Nambak District Hospital, Luang Prabang, Laos

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Moser W, Sayasone S, Xayavong S, Bounheuang B, Puchkov M, Huwyler J, Hattendorf J, Keiser J. Efficacy and tolerability of triple drug therapy with albendazole, pyrantel pamoate, and oxantel pamoate compared with albendazole plus oxantel pamoate, pyrantel pamoate plus oxantel pamoate, and mebendazole plus pyrantel pamoate and oxantel pamoate against hookworm infections in school-aged children in Laos: a randomised, single-blind trial. Lancet Infect Dis. 2018 Jul;18(7):729-737. doi: 10.1016/S1473-3099(18)30220-2. Epub 2018 Apr 16. PMID 29673735